CLINICAL TRIAL: NCT03970265
Title: Development of a Method to Extract Interstitial Lung Fluid and Epithelial Lining Fluid for Antibiotic Concentration Measurement in Explanted Lung Tissue (Feasibility Study)
Brief Title: Development a Method to Extract Antibiotic Concentration From Interstitial Lung and Epithelial Lining Fluid.
Acronym: ALF
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Michael Zoller MD, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: LMU 18-928
Record Dates: First submitted 2019-05-27; First posted 2019-05-31 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Lung Transplantation
Keywords: Interstitial lung fluid; Epithelial lining fluid; Antibiotic concentration in the lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: extraction of ELF and ILF from explanted lung tissue; meropenem concentration in ELF and ILF; ELF on postoperative day 1-5 when bronchoscopy is performed within clinical routine. — Interventions will only be performed on explanted lung tissue ex vivo and on supernatant of bronchoscopy and are therefore non-invasive

SUMMARY:
Infections are critical factors for the survival of critically ill patients. A serious problem is the high variability of antibiotic concentrations in critically ill patients. This may result in the risk of underdosage with possible ineffective therapeutic levels as well as in the risk of overdosage with possible adverse and toxic effects. Essential for the effectiveness of antibiotic therapy is the antibiotic concentration at target site. The goal of this study is to establish a method to extract Interstitial Lung Fluid (ILF) and Epithelial Lining Fluid (ELF) for antibiotic concentration measurements in patients following lung Transplantation and to calculate a tissue/serum concentration ratio. Improved knowledge regarding tissue penetration of Antibiotics may help to optimize drug dosing and management.

DETAILED DESCRIPTION:
Informed consent will be obtained prior to inclusion. 30 patients following lung Transplantation at the University Hospital of Munich will be included in this study. Intravenous Meropenem will be administered as perioperative antibiotic prophylaxis for lung transplantation. Interstitial Lung Fluid and Epithelial Lining Fluid will be extracted immediately after explantation of the lung from explanted lung tissue. Concentrations of antibiotics will be determined by liquid chromatography-mass spectrometry (LC-MS/MS) in ILF and ELF. Serum samples will be collected according to our in clinical routine established therapeutic drug monitoring. Tissue/Serum concentration ratio will be calculated. ELF will be collected on postoperative day 1-5 when bronchoscopy is performed during clinical routine. Numerous clinical and laboratory parameters will be determined. The investigators expect that correlations between antibiotic target site and blood concentrations and clinical and laboratory parameters will be found.

ELIGIBILITY:
Inclusion Criteria:

1. Lung Transplantation at University Hospital of Munich
2. Administration of Meropenem as perioperative antibiotic prophylaxis
3. Valid informed consent subscribed by the patient prior to inclusion

Exclusion Criteria:

1. missing informed consent
2. subsequent withdrawal of the participation in the study by the patient or the guardian

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant patients at University Hospital of Munich
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Meropenem concentration in Interstitial Lung Fluid (ILF) and Epithelial Lining Fluid (ELF) in 30 explanted lungs | 1 year
  The primary goal of this study is to measure Meropenem concentration by LC-MS/MS in ELF and ILF from 30 explanted lung tissue.

SECONDARY OUTCOMES:
Correlation of blood and tissue concentrations of Meropenem | 1 year
  Calculation of tissue/serum concentration ratio will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zoller, Dr.med., Principal Investigator — Department of Anaesthesiology, University Hospital, LMU Munich; Ines Schroeder, Dr.med., Principal Investigator — Department of Anaesthesiology, University Hospital, LMU Munich; Mathias Brügel, Dr.med., Principal Investigator — Institute of Laboratory Medicine, University Hospital, LMU Munich; Michael Vogeser, Prof.Dr.med., Study Chair — Institute of Laboratory Medicine, University Hospital, LMU Munich; Christina Scharf, Dr.med., Study Chair — Department of Anaesthesiology, University Hospital, LMU Munich; Uwe Liebchen, Dr.med., Study Chair — Department of Anaesthesiology, University Hospital, LMU Munich; Eike Speck, Dr.med., Study Chair — Department of Anaesthesiology of the University Hospital of Munich; Paal Michael, Dr.rer.nat., Study Chair — Institute of Laboratory Medicine of the University Hospital of Munich; Alexander Indrich, Dr.med., Study Chair — Department of Anaesthesiology of the University Hospital of Munich; Daniel Siegl, Dr.med., Study Chair — Department of Anaesthesiology of the University Hospital of Munich; Bernhard Zwissler, Prof.Dr.med, Study Director — Department of Anaesthesiology of the University Hospital of Munich; Daniel Teupser, Prof.Dr.med., Study Director — Institute of Laboratory Medicine of the University Hospital of Munich
Locations (1):
- Department of Anaesthesiology of the University Hospital of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paal M, Scharf C, Denninger AK, Ilia L, Kloft C, Kneidinger N, Liebchen U, Michel S, Schneider C, Schropf S, Schuster C, Vogeser M, Weinelt F, Zander J, Zoller M, Schroeder I. Target Site Pharmacokinetics of Meropenem: Measurement in Human Explanted Lung Tissue by Bronchoalveolar Lavage, Microdialysis, and Homogenized Lung Tissue. Antimicrob Agents Chemother. 2021 Nov 17;65(12):e0156421. doi: 10.1128/AAC.01564-21. Epub 2021 Sep 27. PMID 34570645